CLINICAL TRIAL: NCT03874494
Title: A Phase III, Multicenter, Randomized, Double-blind, Active-Controlled Study (Aripiprazole Tablets) to Evaluate the Efficacy and Safety of Brexpiprazole in the Treatment of Adults With Acute Schizophrenia
Brief Title: Safety and Efficacy of Brexpiprazole in the Treatment of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-403-00027
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Brexpiprazole; Non-inferiority
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brexpiprazole (Experimental): 2-4 mg/day, once daily for 6 weeks, oral administration
  Interventions: Drug: Brexpiprazole
- Aripiprazole (Active Comparator): 10-20 mg/day, once daily for 6 weeks, oral administration
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole 2-4 mg/day
  Other Names: Brexpiprazole Tablets
  Arms: Brexpiprazole
Drug: Aripiprazole — Aripiprazole 10-20 mg/day
  Other Names: Aripiprazole Tablets
  Arms: Aripiprazole

SUMMARY:
This study is a phase III, multicenter, randomized, double-blind, active-controlled, non-inferiority trial designed to assess the efficacy and safety of Brexpiprazole in the Treatment of Adults With Acute Schizophrenia. A total of approximately 370 subjects will be included in the study, and randomized to Brexpiprazole (2~4 mg/d) or Aripiprazole (10~20 mg/d) in a 1:1 ratio.

DETAILED DESCRIPTION:
Screening Phase: It will begin when informed consent form (ICF) is signed and be a maximum of 14 days, to evaluate the inclusion/exclusion criteria, collect information such as demographic data, medical history, wash out previous antipsychotic agents and other prohibited concomitant medications.

Double-blind Treatment Phase: It lasts 6 weeks; the purpose is to compare the efficacy and safety of Brexpiprazole with Aripiprazole in the treatment of adults with acute schizophrenia.

Follow-up Phase: All subjects will be followed up for safety reasons via telephone contact or clinic visit 30 (+ 2) days after the last dose of investigational medicinal product, collecting safety information (adverse events and concomitant medication).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent form by subjects and subject's legal guardian or legally acceptable representative.
2. The subjects and subject's legal guardian or legally acceptable representative have the ability to understand the nature of the trial, agree to comply with the prescribed medication and dosage regimens, complete the scheduled visits, report the adverse events and concomitant medication to investigators, and to be reliably rated on psychiatrically scales.
3. At the time of signing informed consent, 18 ≤ age of the subject ≤ 65.
4. Subjects who are diagnosed with schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by Mini International Neuropsychiatric Interview (MINI).
5. Subjects who are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by meeting ALL of the following criteria at the screening and baseline visit:

   ● PANSS total score ≥ 70;
   * Score ≥ 4 on at least 2 of the following PANSS items :

   ( P2 Conceptual disorganization, P3 Hallucinatory behavior, P6 Suspiciousness / persecution, G9 Unusual thought content ) ● CGI-S score ≥ 4;
6. Subjects willing to discontinue all prohibited psychotropic medications to meet protocol-required washouts prior to and during the trial period.

Exclusion Criteria:

1. From ICF to 30 days after the last dose, females of childbearing potential and male subjects who are not willing or cannot practice contraceptive methods.
2. Females who are pregnant or breastfeeding.
3. Subjects who have been hospitalized for > 21 days for the current acute episode at the time of the Baseline visit, excluding hospitalization for psychosocial reasons.
4. Subjects with improvement of ≥ 30% in total PANSS score between the screening and baseline assessment. Improvement in PANSS score= (score at screening-score at baseline)/ (score at screening-30)*100%.
5. Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history of failure to respond to 2 adequate different antipsychotic medications with a minimum of 6 weeks at clinically efficacious tolerated doses. Subjects who have a systemic treatment of clozapine.
6. Subjects with a current DSM-IV-TR Axis I diagnosis (including but not limited to): schizoaffective disorder, MDD, bipolar disorder, post-traumatic stress disorder, anxiety disorders, delirium, dementia, amnestic or other cognitive disorders.
7. Subjects with a current DSM-IV-TR Axis II diagnosis: borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorders.
8. Subjects who present a serious risk of suicide:

   ● Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 or 5 and meeting the criteria for this C-SSRS Item 4 or 5 occurred within the last 6 months; OR

   ● Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items and meeting the criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years; OR

   ● Subjects who, in the opinion of the investigator, present a serious risk of suicide
9. Subjects with clinically diagnosed tardive dyskinesia, as determined by a score of ≥ 3 in Item 8 of the AIMS at the Screening visit.
10. Subjects with a score of 5 in the BARS global clinical assessment of akathisia at Screening or Baseline.
11. Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the 180 days prior to Screening Visit; including alcohol and benzodiazepines, but excluding caffeine and nicotine.
12. Subjects with uncontrolled thyroid disease and/or abnormal free thyroxine (FT4) examination results at Screening, unless it has been confirmed by the investigator that the condition has been stabilized by medication > 90 days before screening
13. Subjects with type I diabetes or uncontrolled type II diabetes. Subjects with type II diabetes may be eligible for the trial if their condition is stable as determined by satisfying ALL of the following criteria:

    * HbA1c < 7.0%, AND
    * Glucose must be ≤ 125 mg/dL or ≤ 6.94 mmol/L (fasting) or < 200 mg/dL or < 11.1 mmol/L (non-fasting) at Screening. If the non-fasting glucose is ≥ 200 mg/dL or ≥ 11.1 mmol/L, subjects must be retested in a fasted state and the retest value must be ≤ 125 mg/dL or ≤ 6.94 mmol/L, AND
    * Subjects have maintained a stable regimen of oral anti-diabetic medication(s) for at least 28 days prior to screening or diabetes has been well-controlled by diet for at least 28 days prior to screening, AND
    * Subjects have not had any hospitalizations within the 12 months prior to screening due to diabetes or complications related to diabetes, AND
    * Subjects whose diabetes is not newly diagnosed during screening for the trial.
14. Subjects with uncontrolled hypertension (diastolic blood pressure > 95 mmHg in any position) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in systolic blood pressure and/or a decrease of ≥ 20 mmHg in diastolic blood pressure after at least 3 minutes standing compared to the previous supine blood pressure, OR development of symptoms.
15. Subjects with a history of ischemic heart disease or history of myocardial infarction, congestive heart failure (whether controlled or uncontrolled), angioplasty, stenting, or coronary artery bypass surgery.
16. Subjects who have a history or severe organic disease of vital organs (including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease).
17. Subjects with epilepsy or a history of seizures, except for a single seizure episode, for instance childhood febrile seizure and post traumatic or alcohol withdrawal.
18. The following laboratory test and ECG results are exclusionary:

1) Platelets ≤ 75,000/mm3 (≤ 75 x 109 /L) 2) Hemoglobin ≤ 9 g/dL (90 g/L) 3) Neutrophils ≤ 1,000/mm3 (1 x 109 /L) 4) AST or ALT > 2 × ULN 5) CPK > 3 × ULN 6) Creatinine ≥ 2 mg/dL (176.8 µmol/L) 7) HbA1c ≥ 7.0% 8) QTc ≥ 450 msec (for males) or ≥ 470 msec (for females) in ECG 19. Subjects who received ECT within 60 days of screening. 20. Subjects with a history of neuroleptic malignant syndrome (NMS). 21. Subjects with a history of true allergic response (ie, not intolerance) to more than one class of medications.

22. Subjects who participated in a clinical trial within the last 90 days or who participated in two or more clinical trials within the past year.

23. Any subject who, in the opinion of the investigator, should not participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) total score | 6 weeks
  The Positive and Negative Syndrome Scale (PANSS) measures psychotic symptoms in patients with schizophrenia. PANSS includes 30 items (7 items for positive symptoms, 7 items for negative symptoms, and 16 items for general psychopathology symptoms), and each item ranges from 1 to 7. The PANSS total score is a sum of scores from all items, ranging from 30 to 210, where a higher score represents severer psychotic symptoms in patients with schizophrenia.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) score | 6 weeks
  The Clinical Global Impression-Severity (CGI-S) score ranges from 1 to 7. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
The Personal and Social Performance Scale (PSP) global score | 6 weeks
  The Personal and Social Performance Scale (PSP) contains four domains: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. A higher domain score represents worse functional performance in each domain. The final global score is defined according to a summary instruction table converting four domain scores into a single, overall rating from 1 to 100, where a higher score represents better personal and social function.
Positive and Negative Syndrome Scale (PANSS) positive scale score | 6 weeks
  The Positive and Negative Syndrome Scale (PANSS) positive scale includes 7 items, assessing positive symptoms in schizophrenia such as delusion, hallucinatory or excitement, and each item ranges from 1 to 7. The positive scale score is a sum of scores from the 7 items, ranging from 7 to 49, where a higher score represents severer schizophrenia positive symptoms.
Positive and Negative Syndrome Scale (PANSS) negative scale score | 6 weeks
  The Positive and Negative Syndrome Scale (PANSS) negative scale includes 7 items, assessing negative symptoms in schizophrenia such as blunted affect or emotional withdrawal, and each item ranges from 1 to 7. The negative scale score is a sum of scores from the 7 items, ranging from 7 to 49, where a higher score represents severer schizophrenia negative symptoms.
Clinical Global Impression-Improvement (CGI-I) score | 6 weeks
  The Clinical Global Impression-Improvement (CGI-I) score ranges from 1 to 7. A higher score represents a poorer clinical impression on the patient's improvement based on investigator/clinician's judgment.
Response rate | 6 weeks
  defined as reduction of ≥ 30% from baseline in PANSS Total Score OR CGI-I score of 1 [very much improved] or 2 [much improved]) at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Zhang, PhD, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- No.15 Yanyin Road, Yanta District, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No